CLINICAL TRIAL: NCT06082479
Title: The Effect of Cryotherapy on Pain and Substancs P Level in Patients With Symptomatic Apical Periodontitis (A Randomized Clinical Trial)
Brief Title: The Effect of Intra Oral Cryotherapy in Patients With Symptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maram Obeid, Professor of Endodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 304
Record Dates: First submitted 2023-09-29; First posted 2023-10-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Post Operative Pain; Inflammation
Keywords: Cryotherapy; substance P; apical periodontitis; post operative pain
MeSH Terms: conditions — Pain, Postoperative; Inflammation; Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: This study was designed to be a randomized, controlled, single-blinded, single-center clinical trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A) Sequence generation;was done using a random sequence number generated by computer software.
  B) Allocation Concealment Mechanism: Folded, numbered papers were placed in tightly sealed envelopes containing the patient's coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no application of any type of cryotherapy.
- cryotherapy group (Active Comparator): after the completion of the mechanical preparation. A 2.5 x5 centimetre gel pack was placed in the mouth on the vestibular surface of the treated tooth.
  Interventions: Procedure: intraoral cryotherapy,ice gel

INTERVENTIONS:
Procedure: intraoral cryotherapy,ice gel — A cold pack (ice gel enveloped by a sealed plastic cover) measuring 2.5 x 5 centimetres was placed intraorally on the vestibular surface of the treated tooth. Each cold pack was kept for ten minutes.3 packs were used for each patient, for a total time of 30 minutes.Patients were instructed to remove the cold pack for 1-2 minutes if they felt extreme cold or a burning sensation .The temperature of the gel was checked by a digital thermometer (Brannan, UK) after it was removed from the freezer and kept in an ice box (Cosmoplast, UAE) containing a cooling gel (Exam Packaging, Belgium).
  Other Names: cold therapy,ice pack
  Arms: cryotherapy group

SUMMARY:
The participants were divided into two groups: Group I (cryotherapy) (n =10) after the completion of the mechanical preparation intra oral cryotherapy was applied. Group II (control) (n =10) received standard root canal treatment without the application of any type of cryotherapy.

DETAILED DESCRIPTION:
1-Patients selection: 20 patients with symptomatic apical peridontitis related to mandibular premolars were selected . After proper anestehsia, Access cavity preparation was performed. The working length measured using apex locator. chemicomechanical preparation was done. for cryotherapy group: cold pack (ice gel enveloped by a sealed plastic cover) measuring 2.5 x 5 centimetres was placed intraorally on the vestibular surface of the treated tooth for a total time of 30 minutes. apical fluid sample was collected by paper point and the root canal was then filled using gutta percha and resin-based sealer.The access cavity was sealed using glass ionomer restoration. for the control group normal treatment was done and apical fluid was collested also before obturation.

ELIGIBILITY:
Inclusion criteria:

* clinical diagnosis of symptomatic apical periodontitis related to ving a mandibular single-rooted premolars
* radigraphically: absence of periapical radiolucency on x ray.

Exclusion criteria:

* The presence of any systemic disease or allergic reactions
* Vulnerable population: prisoners, pregnant women, mentally ill people, etc.
* Use of analgesic or antibiotic medication within three days
* A radiographically untraceable canal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Level of post operative pain using 10 cm visual analoge scale (VAS) | after 6hours, 24hours, 48hours, 72hours h, and 7days after the visit
  On a10-cm Visual Analogue Scale (VAS) questionnaire, each patient reported their level of pain as follows: There is no pain at 0, 1-3, mild, 4-6, moderate, 7-9, severe, and 10, the worst pain.

SECONDARY OUTCOMES:
Level of inflammatory mediator substance P in apical fluid | base line: immediately after procedure.the second is 30 minutes later in both groups.
  Apical fluid samples were obtained using paper points size 25 passing 2 mm beyond the apex.where they were soaked by the periapical interstitial fluid for 1 minute .Four mm from the tip of each paper point was cut and dropped into 1.5-mL Eppendorf tubes (Swanscombe, UK) with 1 mL (pH 7.4) phosphate buffered saline, then stored at -80°C. Levels of substance p were measured using the ELISAtest.

CONTACTS AND LOCATIONS:
Overall Officials: Maram F Obeid, Professor, Study Director — Faculty of Dentistry,Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
detailed Statistical Analysis Plan
Supporting Information: SAP
Time Frame: 2025 ,available for a year
Access Criteria: review the purpose of request

REFERENCES:
- [Background] Gundogdu EC, Arslan H. Effects of Various Cryotherapy Applications on Postoperative Pain in Molar Teeth with Symptomatic Apical Periodontitis: A Preliminary Randomized Prospective Clinical Trial. J Endod. 2018 Mar;44(3):349-354. doi: 10.1016/j.joen.2017.11.002. Epub 2018 Feb 3. PMID 29398090
- [Background] Keskin C, Aksoy A, Kalyoncuoglu E, Keles A, Ilik AA, Komec O, Yuzgulec E, Akgun H, Alak SG, Tokur O. Effect of intracanal cryotherapy on the inflammatory cytokine, proteolytic enzyme levels and post-operative pain in teeth with asymptomatic apical periodontitis: A randomized clinical trial. Int Endod J. 2023 Aug;56(8):932-942. doi: 10.1111/iej.13937. Epub 2023 May 30. PMID 37222468
- See also: worked on inflammatory mediators in similar matter — https://dsu.journals.ekb.eg/article_192084.html